CLINICAL TRIAL: NCT06101264
Title: Application of Virtual Reality in Post-Operative Recovery of a Pediatric Scoliosis Patient Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Connecticut Children's Medical Center (Other)
Collaborators: University of Connecticut (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-064-CCMC
Record Dates: First submitted 2023-10-16; First posted 2023-10-26 (Actual); Results first posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Adolescent Idiopathic Scoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Virtual Reality (Experimental): Participants will receive a post-operative virtual reality intervention following corrective surgery for idiopathic scoliosis.
  Interventions: Device: Virtual Reality
- Control (Experimental): Patients not receiving virtual reality intervention following corrective surgery for idiopathic scoliosis.
  Interventions: Device: Control

INTERVENTIONS:
Device: Control — Control patients following spinal fusion for adolescent idiopathic scoliosis that receive no virtual reality sessions.
  Arms: Control
Device: Virtual Reality — Patients will undergo a 20 minute virtual reality session prior to each physical therapy session following spinal fusion for adolescent idiopathic scoliosis. Virtual reality sessions will continue until functionally cleared by physical therapy.
  Arms: Virtual Reality

SUMMARY:
The purpose of this study is to assess the effect of virtual reality on subjective post-operative pain, total inpatient narcotic administration, and mobilization with physical therapy in pediatric patients who have undergone surgical correction for idiopathic scoliosis.

DETAILED DESCRIPTION:
All pediatric patients (ages 13-18) at Connecticut Children's Medical Center undergoing corrective scoliosis surgery for idiopathic scoliosis are eligible and will be approached for consent and inclusion into the study. This is a prospective pilot study, and all enrolled patients will receive a virtual reality (VR) intervention using a commercially available device manufactured by Oculus. The VR software will simulate a low physical load environment, such as an underwater space exploration game. Starting on postoperative day 1, the prospective cohort will undergo a 20-minute VR session 30 minutes prior to each physical therapy session. There will be two physical therapy sessions scheduled daily for the participant. Outcome measures will be assessed before and after the VR session and after the physical therapy session. The following procedures will continue daily until the participant is cleared for hospital discharge. Patients that met study eligibility but elected not to participate in the VR intervention were analyzed as the control group.

ELIGIBILITY:
Inclusion Criteria:

* All pediatric patients (ages 13-18) at Connecticut Children's undergoing surgical correction for idiopathic scoliosis over a span of 12 months

Exclusion Criteria:

* History of seizures
* Cognitive developmental delay precluding participation in VR
* Head or neck surgery that does not allow a head-mounted display to be worn safely
* Chronic pain requiring the daily use of opioids for more than 2 weeks prior to the procedure
* Non-English speakers
* Side effects during screening
* Patients with vagal nerve stimulators, cardiac pacemakers, and/or cochlear implants that may receive interference from the VR device

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Hersh, MD, Principal Investigator — Connecticut Children's Medical Center
Locations (1):
- Connecticut Children's Medical Center, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Virtual Reality Intervention: Participants will receive a post-operative virtual reality intervention following corrective surgery for idiopathic scoliosis.
  Virtual Reality Intervention: Participants will be given a virtual reality (VR) intervention following corrective scoliosis surgery for adolescent idiopathic scoliosis. The VR intervention will utilize a commercial device manufactured by Oculus. The intervention will utilize a software that simulates a low-physical load environment for the user. Starting on postoperative day 1, the participant will receive a 20-minute VR intervention 30 minutes prior to each physical therapy session. There will be two physical therapy sessions daily. Outcome measures will be assessed before and after every VR intervention and after the physical therapy session. The VR interventions will continue for each postoperative day until the participant is discharged from the hospital.
- Control: Patients that underwent spinal fusion for adolescent idiopathic scoliosis but did not receive virtual reality interventions.
Period: Overall Study
Arm/Group | Virtual Reality Intervention | Control
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control: Control: A retrospective chart review was performed to identify patients that met inclusion criteria. These patients did not undergo virtual reality intervention however the standard of care was identical in both groups. Outcome measures will be assessed before and after the physical therapy session
- Total: Total of all reporting groups
Arm/Group | Virtual Reality Intervention | Control | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.1 (1.6) | 15.8 (1.3) | 15.5 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 3 | 12
  Male | 1 | 7 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 8 | 3 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Average Change in Subjective Pain Level Using a 10 Point Likert Scale
Description: This tool uses a 10-point scale that ranges from 0 (no pain) to 10 (worst possible pain). Pain will be assessed using this tool before and after every physical therapy session. The change in pain before and after each physical therapy session will be calculated and averaged across each patient.
Time Frame: 2 times daily postoperatively until hospital discharge (up to 60 days postoperatively)
Measure: Mean (Standard Deviation); unit: pain score
Groups:
- Control: Control: A retrospective chart review was performed to identify patients that met inclusion criteria. These patients did not undergo virtual reality intervention however the standard of care was identical in both groups. Outcome measures will be assessed before and after the physical therapy session,
Arm/Group | Virtual Reality Intervention | Control
Number analyzed (Participants) | 10 | 10
pain score | -0.72 (1.2) | 0.61 (1.1)

2. Secondary Outcome: Total Amount of Administered Opioids During the Post-operative Period
Description: Opioid utilization will be assessed by calculating the total inpatient dose of opioids administered (as documented in the electronic medical record) during the post-operative period, starting from post-operative day 1 until hospital discharge.
Time Frame: From post-operative day 1 until hospital discharge (up to 60 days postoperatively)
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Virtual Reality Intervention | Control
Number analyzed (Participants) | 10 | 10
mg | 55.7 (31.7) | 49.9 (19.1)

3. Secondary Outcome: Average Number of Physical Therapy Sessions Prior to Receiving Clearance by Physical Therapy Staff
Description: In the postoperative stage, each participant will receive two physical therapy sessions daily. Physical therapy sessions will continue daily until the participant is given clearance by the physical therapy team. To assess the mobilization of participants postoperatively, the total number of physical therapy sessions the participants attend prior to receiving clearance will be noted. The number of total attended physical therapy sessions during the postoperative stage will be averaged across all participants.
Time Frame: Post-operative day 1 until clearance by physical staff (up to 60 days postoperatively)
Measure: Mean (Standard Deviation); unit: sessions
Arm/Group | Virtual Reality Intervention | Control
Number analyzed (Participants) | 10 | 10
sessions | 3.2 (1.7) | 3.2 (1.1)

ADVERSE EVENTS:
Time Frame: Adverse effects were collected during the virtual reality sessions until the patient was discharged from the hospital, up to 60 days postoperatively.
Groups:
- Control: Patients that underwent corrective surgery for idiopathic scoliosis but did not undergo virtual reality sessions.
Arm/Group | Virtual Reality Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 6/10 | 0/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Virtual Reality Intervention (N=10) | Control (N=10)
Fatigue (General disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 3 | 0
Headache (Nervous system disorders) | 2 | 0
Eye Strain (Eye disorders) | 2 | 0
Dizziness (Nervous system disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
This study allocation of patients to the control group if they declined participation in the virtual reality sessions and is such not a true randomized controlled trial. Further, our prospective study has a small sample size as it is intended as a pilot study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-12): https://cdn.clinicaltrials.gov/large-docs/64/NCT06101264/Prot_SAP_000.pdf